CLINICAL TRIAL: NCT04746261
Title: A Randomized Clinical Study of "Attempted Suicide Short Intervention Program" in Swedish Healthcare - ASSIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-02360
Record Dates: First submitted 2020-08-12; First posted 2021-02-09 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Suicide, Attempted
MeSH Terms: conditions — Suicide, Attempted | interventions — Therapeutics; Patient Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASSIP plus treatment as usual (Experimental): ASSIP according to manual. Treatment as usual will be multidisciplinary and combine psychotherapy, pharmacotherapy and other treatments as well as referral to specialist psychiatry or primary care as required.
  Interventions: Behavioral: ASSIP + treatment as usual; Other: Treatment as usual and patient safety
- Treatment as usual (Active Comparator): Treatment as usual will be multidisciplinary and combine psychotherapy, pharmacotherapy and other treatments as well as referral to specialist psychiatry or primary care as required.
  Interventions: Other: Treatment as usual and patient safety

INTERVENTIONS:
Behavioral: ASSIP + treatment as usual — ASSIP:
  First session: Videotaped narrative interview focusing on the background to the suicidal crisis.
  Second session: Video playback. The patient and the therapist watch the recorded interview together, stopping the film regularly to add information. The patient is given a psychoeducational text to read and comment on as homework.
  Third session: Compilation of a written case formulation of the individual's vulnerability and triggering events that preceded the suicidal crisis. Individual preventive measures are developed by the patient and the therapist together and written down in a document that the patient keeps and which is attached to the patient's medical record.
  Fourth session (optional): Mini-exposure.
  Standardized letters: The therapist contacts the patient by letter during two years, every three months the first year and every six months the second year.
  Treatment as usual: As described bellow
  Arms: ASSIP plus treatment as usual
Other: Treatment as usual and patient safety — All patients follow their usual care, regardless of whether they are treated with ASSIP or not. Usual care is multidisciplinary and combines psychotherapy, pharmacotherapy and other treatments, including referral to specialist psychiatric units or primary care. This depends on the assessments made by the patient's usual care provider. Treatment as usual is monitored by the research team through a standardised medical record review.
  In order to increase patient safety, some standardisation of usual care takes place. The research nurse communicates with the referring healthcare provider to ensure that the patient receives a follow-up appointment within the usual care setting after the initial visit and the research team informs the usual care provider and acts when acute suicide risk is detected. In most sites, some information from SIS, CSSR-S and MINI assessments is noted in the patient's medical records.

SUMMARY:
This is a randomized study of ASSIP as a treatment for patients who have recently made a suicide attempt. Six psychiatric clinics from four regions in Sweden are included. Together 460 patients will be recruited. Patients will be randomized to ASSIP as a supplement to treatment as usual or to treatment as usual only.

The overall aim of the study is to evaluate whether ASSIP, a short-term clinical intervention, can prevent future suicidal behavior in people who have attempted suicide better than just conventional treatment. The project also investigates whether there are any specific factors that may be related to ASSIP's potential effectiveness and whether ASSIP has health economic benefits.

Only patients who give their written consent will be included in the study. Those who meet the inclusion and no exclusion criteria at screening / visit 1 undergo an assessment according to an interview protocol, self-assessment form, and self-assessment scales. Thereafter, the patient is randomized via an electronic system to either ASSIP plus standard treatment or only standard treatment. All patients, regardless of which treatment they are randomized to, will be followed up for two years with a telephone interview and self-assessment scales month 3, 12 and 24. Data from medical records and registers will also be collected.

DETAILED DESCRIPTION:
Purpose and aims:

The overall purpose of this project is to evaluate ASSIP for the prevention of future suicidal behavior in persons who attempt suicide. The specific goals are a) to examine the effectiveness of Attempted Suicide Short Intervention Program (ASSIP) in reducing new suicide attempts in Swedish healthcare, b) to identify factors associated with the effectiveness of ASSIP, c) to construct a cost-effectiveness model of ASSIP.

Background:

According to a consensus position paper from the evidence-based national suicide prevention task force in Europe, health care approaches with high evidence include treatment of depression and ensuring chain of care. These strategies are in line with Swedish guidelines. However, several recent international studies suggest that interventions specifically targeted to prevent suicide attempts may be more successful and that brief psychological interventions are of interest . One promising brief psychotherapeutic intervention to prevent new suicide attempts in suicide attempters is ASSIP . An RCT from Switzerland that included 120 patients showed an 80% risk reduction for new suicide attempt within two years, when ASSIP was added on to treatment as usual (TAU) compared to TAU alone.

Study design:

This is an evaluator-blinded, multicenter randomized controlled trial (RCT). The patients will be examined with a structured interview and self-rating scales at baseline (first visit), and structured telephone interviews, self-rating scales and medical record screening at 3 months, 12 months and 24 months follow up. Completed suicides will be detected through the Cause of Death Register. The study will also collect information from the National Board of Health and Welfare (NBHW), National Prescribed Drugs Register (NPDR), Longitudinal integrated database for health insurance and labour market studies (LISA) and the Swedish Social Insurance Agency (Försäkringskassan).

Randomization: After the first visit, the patients will be randomized to ASSIP+ TAU or TAU only, using stratified randomization according to clinical site. The randomization will be performed through REDCAP, a web-based application for electronic data collection in research studies. Expected site differences: To map the variation of TAU with site, age, gender, ICD diagnoses and previous suicide attempts, health care contacts and treatments a TAU check list will be used.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Signed informed consent to participate in the study.
* Contact with psychiatric health care after a suicide attempt within 3 months before the baseline visit
* Booked meeting or visit in psychiatry or primary care after visit 1

Exclusion Criteria:

* Psychotic illness with current delusions, hallucinations or other negative symptoms that may affect the therapy.
* Known emotionally unstable personality disorder (ICD 10) noted in the medical record
* Inability to undergo therapy without an interpreter
* Mental retardation, dementia, or other circumstances that make it difficult to understand the meaning of participating in the study and giving informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of suicide attempts up to 24 months after inclusion | 24 months after inclusion in study
  Repeated telephone follow up at 3, 12 and 24 months after inclusion. Medical records data. Register data
Number of suicide attempts up to 12 months after inclusion | 12 months after inclusion in study
  Repeated telephone follow up at 3, 12 after inclusion. Medical records data. Register data.
Number of suicide attempts up to 3 months after inclusion | 3 months after inclusion in study
  Telephone follow up at 3 months after inclusion. Medical records data. Register data.
Incremental Cost-Effectiveness Ratio( ICER). | 24 months after inclusion
  RCT outcomes put into perspective using a health-economic model with a life-time horizon, evidence from literature and complementary register data.

SECONDARY OUTCOMES:
Number of suicidal thoughts/plans within 24 months after inclusion | 24 months after inclusion in study
  Repeated self ratings, suicidal thoughts defined as MADRS-S (Montgomery-Asberg Depression Rating Scale) question 9 score above or equal to 4 at 3, 12 and 24 months
Number of suicidal thoughts/plans within 12 months after inclusion | 12 months after inclusion in study
  Repeated self ratings, suicidal thoughts defined as MADRS-S (Montgomery-Asberg Depression Rating Scale) question 9 score above or equal to 4 at 3 and 12 months
Number of suicidal thoughts/plans within 3 months after inclusion | 3 months after inclusion in study
  Repeated self ratings, suicidal thoughts defined as MADRS-S (Montgomery-Asberg Depression Rating Scale) question 9 score above or equal to 4 at 3 months
Health care contacts and treatments | 24 months after inclusion
  Number and type of healthcare contacts according to telephone interviews and medical records
Changes in Quality of life | 3 months
  Self reported quality of life reported according to the EuroQol Research Foundation, EQ-5D-5L at 3 months follow up in comparison with first visit.The EQ-5D-5L consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: Each dimension has 5 levels: A higher 1-digit number mean a worse outcome. High scores on the EQ VAS mean a better outcome.
Changes in Quality of life | 12 months
  Self reported quality of life reported according to the EuroQol Research Foundation, EQ-5D-5L at 12 months follow up in comparison with first visit.The EQ-5D-5L consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: Each dimension has 5 levels: A higher 1-digit number mean a worse outcome. High scores on the EQ VAS mean a better outcome.
Changes in Quality of life | 24 months
  Self reported quality of life reported according to the EuroQol Research Foundation, EQ-5D-5L at 24 months follow up in comparison with first visit.The EQ-5D-5L consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: Each dimension has 5 levels: A higher 1-digit number mean a worse outcome. High scores on the EQ VAS mean a better outcome.
Periods of employment, unemployment, education, military service or pension | 24 months
  Periods of employment, unemployment, education, military service or pension registered in the Longitudinal integrated database for health insurance and labour market studies (LISA)
Amount of income from employment, social insurance, student aid, pension and unemployment benefits. | 24 months
  Amount of income from employment, social insurance, student aid, pension and unemployment benefits registered in the Longitudinal integrated database for health insurance and labour market studies (LISA)
Number of days with sickness and disability benefits | 24 months
  Number of days with sickness or disability benefits registered according to the Swedish Social Insurance Agency

CONTACTS AND LOCATIONS:
Overall Officials: Åsa Westrin, professor, Principal Investigator — Region Skane
Locations (2):
- Sweden (2):
  - Region Skåne, psykiatri & habilitering, psykiatriforskning skane, Vuxenpsykiatri Lud, Lund
  - Region Skåne, psykiatri & habilitering, psykiatriforskning skane,Vuxenpsykiatri Malmoe, Malmo

REFERENCES:
- [Derived] Lindstrom S, Ehnvall A, Bergqvist E, Waern M, Dahlin M, Westrin A. A study protocol of the effectiveness of the Attempted Suicide Short Intervention Program (ASSIP) for recent suicide attempters: a randomized controlled trial. BMC Psychiatry. 2024 Oct 4;24(1):655. doi: 10.1186/s12888-024-06109-z. PMID 39367366